CLINICAL TRIAL: NCT01959737
Title: Influence of Early SSC of Mothers and Their VLBW Infants on Maternal Sensitivity and Responsiveness, Attachment Patterns and Reactivity of HPA Axis. Molecular Characterization of SSC Influence on Stress Signaling Pathways.
Brief Title: Delivery Room Skin-to-skin Study
Acronym: deisy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Katrin Mehler, MD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-075
Record Dates: First submitted 2013-10-07; First posted 2013-10-10 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Very Low Birthweight Infants; Mother Child Interaction; Preterm Infant
Keywords: reactivity of HPA axis
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- visual contact (No Intervention): After initial assessment/stabilization of the VLBW infant, visual contact of mother and infant is permitted for 5 minutes.
- skin-to-skin contact (Experimental): After initial stabilization mother and preterm infant are cared for skin-to-skin for 60 minuter. SSC is supervised by the attending neonatologist.
  Interventions: Procedure: skin-to.skin-contact

INTERVENTIONS:
Procedure: skin-to.skin-contact — Immediately after initial stabilization/ assessment of the VLBW infant, skin-to-skin contact of mother and infant is initiated and kept up for 60 minutes.
  Arms: skin-to-skin contact

SUMMARY:
The first hours after birth are a sensitive period for promotion of optimal mother-child-interaction and secure attachment. Maternal sensitivity and responsivness are high in the first hours after birth due to high oxytocin levels. Developing optimal mother-child-interaction is more difficult for preterm mothers because mother and child are separated after birth and the preterm infant is not able to show strong signs to promote maternal sensitivity. We hypothesize that promoting skin-to-skin contact of VLBW infants and their mothers for 60 minutes within the first hours after birth improves mother-child-interaction at 5 to 6 months corrected age. We also hypothesize that reactivity of HPA axis and molecular patterns of stress signaling pathways differ in preterm infant with or without SSC after birth.

ELIGIBILITY:
Inclusion Criteria:

* Birthweight <1500g, first child, informed consent

Exclusion Criteria:

* Multiples, malformation

Ages: 10 Minutes to 60 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maternal sensitivity and responsiveness | 4 to 6 moinths corrected age
  Maternal sensitivity and responsiveness are assessed with the "Mannheimer Method" for the analysis of mother child interaction. At the infants corrected age of 4 to 6 months a videotape of the mother changing the infants diapers and playing with the infant is used for analysis.

SECONDARY OUTCOMES:
Reactivity of HPA-axis | 36 to 40 weeks corrected age
  Salivary cortisol assessment before and 20 minutes after heel lance
Molecular characterization of stress signaling pathways | 36 to 40 weeks corrected age
  Genomic expression of the Glucocorticoid receptor (NR3C1), Corticotropin releasing hormon (CRH), Corticotropin releasing hormon receptor 1 (CRHR1), serotonin receptor 1A and 2A, serotonin transporter (slc6a4), vasopressin

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Cologne, Department of Neonatology, Cologne, Germany

REFERENCES:
- [Background] Mehler K, Wendrich D, Kissgen R, Roth B, Oberthuer A, Pillekamp F, Kribs A. Mothers seeing their VLBW infants within 3 h after birth are more likely to establish a secure attachment behavior: evidence of a sensitive period with preterm infants? J Perinatol. 2011 Jun;31(6):404-10. doi: 10.1038/jp.2010.139. Epub 2010 Dec 9. PMID 21151007
- [Derived] Trautmann-Villalba P, Heine E, Kribs A, Mehler K. Does early skin-to-skin contact have a long-term effect on the emotional and behavioral development of very preterm infants? Front Psychol. 2024 Nov 11;15:1484419. doi: 10.3389/fpsyg.2024.1484419. eCollection 2024. PMID 39588126